CLINICAL TRIAL: NCT03077672
Title: Mitochondrial DNA as a Biomarker of Sepsis Severity
Acronym: MBOSS
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other); New York Presbyterian Brooklyn Methodist Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1605017267; R01HL055330 (NIH); P01HL108801 (NIH)
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Sepsis Syndrome; Sepsis; Severe Sepsis; Septic Shock; Infection
Keywords: Mitochondrial DNA; Lactate; Mortality; Emergency Department; Intensive Care Unit; Triage; Organ Dysfunction; Biomarker; Prognosis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Shock, Septic; Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Leukocyte Pellet, Mitochondrial DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NYP-WCM: The NYP-WCM cohort will consist of patients presenting to the NewYork-Presbyterian/Weill Cornell Medicine Emergency Department with suspected sepsis.
- NYP-BMH: The NYP-BMH cohort will consist of patients presenting to the NewYork-Presbyterian Brooklyn Methodist Hospital Emergency Department with suspected sepsis.

SUMMARY:
Mitochondria are organelles (a specialized subunit of a cell) responsible for providing cells with energy. For reasons not yet understood, mitochondria will release their DNA into blood in response to cellular injury or cell death.

With a simple blood draw, investigators can measure the amount of mitochondrial DNA in a patient's blood.

The investigators' hypothesis, is that mitochondrial DNA can be used as a surrogate marker of cellular injury to predict patient outcomes. The investigators intend to test their hypothesis by measuring mitochondrial DNA in adult patients presenting to the Emergency Department with sepsis (a life-threatening condition due to an infection) and observing their hospital course.

DETAILED DESCRIPTION:
Despite the advances of modern medicine, sepsis persists as one of the leading causes of death in the United States and poses a significant burden on U.S. health care, accounting for more than $24 billion of total hospital costs in 2013. The high mortality and cost of treating sepsis at least partially stems from the consequences of delayed diagnosis. Unfortunately, this delay is attributable to the broad clinical manifestations of the syndrome and the absence of a specific test for sepsis.

Realizing this, The Society of Critical Care Medicine and the European Society of Intensive Care Medicine have released guidelines emphasizing the need for diagnostic approaches aimed at the early detection of sepsis. The hope is that early recognition will allow for more aggressive upfront management thereby improving patient outcomes.

In 2013, Nakahira et al showed that circulating cell-free mitochondrial DNA levels are associated with sepsis and mortality in patients admitted to the ICU. In contrast to that study, the purpose here is to determine whether circulating cell-free mitochondrial DNA and other biomarkers are associated with the severity of sepsis and 28-day mortality in patients presenting to the ED with sepsis.

To accomplish this task, the investigators intend to prospectively collect specimens from patients presenting to NYP-Weill Cornell and NYP-Brooklyn Methodist with suspected sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Adults presenting to the Emergency Department with suspected sepsis.

Exclusion Criteria:

* Pregnancy.
* Patients with limitations of care at the time of specimen collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We intend to study patients presenting to the NYP-Weill Cornell Medicine Emergency Department and the NYP-Brooklyn Methodist Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | 60 Days
  All-Cause

SECONDARY OUTCOMES:
Association with severity of illness as determined by qSOFA Score | 3 Days
  qSOFA
Association with severity of illness severity of illness as determined by MEDS Score | 3 Days
  MEDS Score
Association with severity of illness as determined by SOFA Score | 3 Days
  SOFA Score
Need for Supportive Measures | Up to 60 Days
  NIPPV, Mechanical Ventilation, Vasopressors, CVVHD, iNO, ECMO
ICU-Free Days | 28 Days
  Number of days free from ICU Admission
Triage Decision | 3 Days
  If the patient was discharged home or admitted to the floor, a step-down unit, or an ICU

CONTACTS AND LOCATIONS:
Overall Officials: John Harrington, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian/Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, de-identified participant data will be able available to individuals six-months after publication of all data.

REFERENCES:
- [Background] Torio CM, Moore BJ. National Inpatient Hospital Costs: The Most Expensive Conditions by Payer, 2013. 2016 May. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #204. Available from http://www.ncbi.nlm.nih.gov/books/NBK368492/ PMID 27359025
- [Background] Nakahira K, Kyung SY, Rogers AJ, Gazourian L, Youn S, Massaro AF, Quintana C, Osorio JC, Wang Z, Zhao Y, Lawler LA, Christie JD, Meyer NJ, Mc Causland FR, Waikar SS, Waxman AB, Chung RT, Bueno R, Rosas IO, Fredenburgh LE, Baron RM, Christiani DC, Hunninghake GM, Choi AM. Circulating mitochondrial DNA in patients in the ICU as a marker of mortality: derivation and validation. PLoS Med. 2013 Dec;10(12):e1001577; discussion e1001577. doi: 10.1371/journal.pmed.1001577. Epub 2013 Dec 31. PMID 24391478